CLINICAL TRIAL: NCT03068221
Title: Clinical Sciences Research Proposal- The Effect of Physical Exercise on Poly Cystic Ovary Syndrome Overweight Female Adolescents
Brief Title: Clinical Sciences Research Proposal- The Effect of Physical Exercise on PCOS Overweight Female Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0342-16CTIL
Record Dates: First submitted 2017-02-12; First posted 2017-03-01 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Polycystic Ovary Syndrome; Overweight
MeSH Terms: conditions — Polycystic Ovary Syndrome; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Poly Cystic Ovary Syndrome (Active Comparator): anaerobic exercise in overweight patients with PCOS
  Interventions: Other: anaerobic exercise
- non Poly Cystic Ovary Syndrome (Active Comparator): anaerobic exercise in overweight patients without PCOS
  Interventions: Other: anaerobic exercise

INTERVENTIONS:
Other: anaerobic exercise — assessing anaerobic exercise status

SUMMARY:
The Poly Cystic Ovary Syndrome (PCOS), is one of the most common reasons for subfertility, oligomenorrhea and amenorrhea. With the occurrence of 6-20% of the general adult women population. One of the main criteria of this syndrome is a hyper androgenic state.

More than 50% of women who have PCOS are overweight. In the teenage population, PCOS is common in 5-10% of teenage girls. A recent research has shown that elite athlete teenage girls have higher serum androgen levels, especially in anaerobic types of sport.

The purpose of this experiment is to examine the reaction of teenage PCOS overweight girls towards anaerobic exercise. To determine if their hyperandrogenic state is more adapted to excel in anaerobic exercise compared to teenage overweight girls without PCOS.

DETAILED DESCRIPTION:
30 teenage and young adult females, aged 10-25 years old. The minimum hormonal age for inclusion is menarche. Overweight- with a Body Mass Index (BMI) percentage above 85%, divided into 2 groups: 15 girls with diagnosed PCOS, and 15 girls without diagnosed PCOS, without any other medical comorbidities. Followed at the pediatric endocrinology unit.

The 2 groups would participate in 2 anaerobic tests to evaluate their performances. The data received will be used to evaluate their anaerobic attributes, and for comparison between the 2 groups to determine any differences.

The participants will be asked to refrain from any form of physical exercise during the previous day.

After explanation to the patient and his parent and obtaining an informed consent, the participants will start the tests.

The first test is the Repeated Sprint Test: The participant will run a distance of 40 meters, for 6 repetitions. The optimal running time will be calculated, total running time and the Performance Decrement of the run will be calculated.

After that, there will be a 1-1.5 hours resting phase. The second test is the "Wingate Test"- the participants will be instructed to pedal at a maximal pace for 30 seconds on an ergometric bicycle against a resistance adjusted according to their BMI. The Peak Anaerobic Power, the Mean Anaerobic Power and the Fatigue Index will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* post menarche female
* PCOS diagnosis
* overweight- BMI above 85 percent.

Exclusion Criteria:

* inability to complete the physical activity due to health issues
* Thyroid dysfunction (hyper-, hypo-)
* hyperprolactinemia
* congenital adrenal hyperplasia

Ages: 10 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Peak anaerobic power | 30 seconds
  The highest produced power (Watt/Kg) during cycling at maximal speed against a weight based calculated resistance for 30 seconds
Mean anaerobic power | 30 seconds
  The mean produced power (Watt/Kg) during cycling at maximal speed against a weight based calculated resistance for 30 seconds

SECONDARY OUTCOMES:
Total running time (Seconds) for a repeated sprint test. | between 40-120 seconds
  6 repetitions of 40 meter sprint, as fastest as the patient can run

CONTACTS AND LOCATIONS:
Overall Officials: Alon Elikaim, MD, Principal Investigator — Meir Medical Center , Tel Aviv University
Locations (1):
- Meir Medical Center , Tel Aviv University, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No